CLINICAL TRIAL: NCT01601392
Title: Effect of Anodal Versus Cathodal Transcranial Direct Current Stimulation on Stroke Recovery: a Pilot Randomized Controlled Trial
Brief Title: Anodal and Cathodal Transcranial Direct Current Stimulation in Stroke Recovery
Acronym: tDCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dina Hatem Elhammady (Other)
Responsible Party: Sponsor-Investigator, Dina Hatem Elhammady, Clinical Professor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: tDCS in stroke recovery
Record Dates: First submitted 2012-05-11; First posted 2012-05-18 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Stroke
Keywords: Ischemic stroke; direct current stimulation; motor threshold; National institutes of Health Stroke Scale; Barthel index scale; Measurement of motor power improvement
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Transcranial Direct Current Stimulation; salicylhydroxamic acid

ARMS (3):
- Anodal tDCS (Experimental)
  Interventions: Procedure: transcranial direct current stimulation (Anodal)
- Cathodal tDCS (Active Comparator)
  Interventions: Procedure: transcranial direct current stimulation (Cathodal)
- Sham (Sham Comparator)
  Interventions: Procedure: transcranial direct current stimulation (Sham)

INTERVENTIONS:
Procedure: transcranial direct current stimulation (Anodal) — The anodal group will receive tDCS for 25 minutes at 2mA daily for 6 consecutive days on the affected hemisphere.
  Arms: Anodal tDCS
Procedure: transcranial direct current stimulation (Cathodal) — The Cathodal group will receive tDCS for 25 minutes at 2mA daily for 6 consecutive days on the unaffected hemisphere.
  Arms: Cathodal tDCS
Procedure: transcranial direct current stimulation (Sham) — The sham group will receive sham tDCS for 25 minutes daily for 6 consecutive days on the affected hemisphere.
  Arms: Sham

SUMMARY:
The purpose of this study will to compare the long-term effect of anodal versus cathodal transcranial direct current stimulation (tDCS) on motor recovery in subacute stroke patients. Forty patients with subacute ischemic stroke will randomly assigned to one of three groups: Anodal, Cathodal and Sham. Each group will receive tDCS at an intensity of 2mA for 25 minutes daily for 6 consecutive days over the affected (Anodal, Sham) or unaffected (Cathodal) motor cortex. Patients will be assessed with National Institutes of Health Stroke Scale (NIHSS), the Barthel index (BI) and the Medical Research Council (MRC) muscle strength scale at baseline, after end of the 6th tDCS session, and then 1, 2 and 3 months later. Motor cortical excitability will be measured at baseline and after the 6th session in both hemispheres.

ELIGIBILITY:
Inclusion Criteria:

* acute hemiparesis with single thromboembolic non-hemorrhagic infarction documented by magnetic resonance imaging (MRI)
* Accept to participate in the study

Exclusion Criteria:

* extensive infarction (taking all territories of middle cerebral artery)
* severe flaccid hemiplegia
* head injury
* Any other neurological disease other than stroke
* previous administration of tranquilizer
* patients who are unable to give informed consent because of severe aphasia, or cognitive deficit.
* Patients with no motor evoked response recorded from First Dorsal Interosseus (FDI) muscle of the affected hand

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Motor power improvement | 3 Months
  improvement in the motor power of paretic patient as measured in one proximal and one distal muscle group testing in upper (shoulder abduction + hand grip) and lower limbs ( hip flexion + toes dorsiflexion).

SECONDARY OUTCOMES:
Motor cortical excitability | 1 Month
  The difference in the motor cortical excitability (RMT, AMT) before and after tDCS

CONTACTS AND LOCATIONS:
Overall Officials: Eman M Khedr, Professor, Principal Investigator — Assiut University
Locations (1):
- Faculty of Medicine, Assiut University, Asyut, Asyut Governorate, Egypt